CLINICAL TRIAL: NCT02100410
Title: On-Eye Evaluation of Contact Lens Axis Location
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: C-12-061
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Results first posted 2014-05-16 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-04

CONDITIONS: Myopia; Astigmatism; Refractive Error
Keywords: Contact Lens; Toric
MeSH Terms: conditions — Myopia; Astigmatism; Refractive Errors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Iteration 2-87-1 (Experimental): Delefilcon A toric contact lenses T1 and T2 worn contralaterally (1 in each eye) for approximately 30 minutes
  Interventions: Device: Delefilcon A toric contact lens T1; Device: Delefilcon A toric contact lens T2
- Iteration 2-87-2 (Experimental): Delefilcon A toric contact lenses T3 and T4 worn contralaterally (1 in each eye) for approximately 30 minutes
  Interventions: Device: Delefilcon A toric contact lens T3; Device: Delefilcon A toric contact lens T4
- Iteration 2-87-3 (Experimental): Delefilcon A toric contact lenses T5 and T6 worn contralaterally (1 in each eye) for approximately 30 minutes
  Interventions: Device: Delefilcon A toric contact lens T5; Device: Delefilcon A toric contact lens T6

INTERVENTIONS:
Device: Delefilcon A toric contact lens T1 — Iteration 2-87-1 with embossed mark
  Arms: Iteration 2-87-1
Device: Delefilcon A toric contact lens T2 — Iteration 2-87-1 without embossed mark
  Arms: Iteration 2-87-1
Device: Delefilcon A toric contact lens T3 — Iteration 2-87-2 with embossed mark
  Arms: Iteration 2-87-2
Device: Delefilcon A toric contact lens T4 — Iteration 2-87-2 without embossed mark
  Arms: Iteration 2-87-2
Device: Delefilcon A toric contact lens T5 — Iteration 2-87-3 with embossed mark
  Arms: Iteration 2-87-3
Device: Delefilcon A toric contact lens T6 — Iteration 2-87-3 without embossed mark
  Arms: Iteration 2-87-3

SUMMARY:
The purpose of this study was to evaluate the axis location of toric contact lenses after 3 minutes of wear. During this 1-visit study, each participant wore 3 pairs of study lenses of various design iterations (2-87-1, 2-87-2, 2-87-3) for an exposure time of approximately 30 minutes each. Each pair consisted of lenses of the same design iteration, 1 lens with embossed mark [TEST1 (T1), TEST3 (T3), TEST5 (T5)], worn on the right eye, and 1 lens without embossed mark [TEST2 (T2), TEST4 (T4), and TEST6 (T6)] worn on the left eye.

ELIGIBILITY:
Inclusion Criteria:

* Sign written Informed Consent.
* Best corrected distance visual acuity greater than or equal to 20/25 in each eye.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* History of any ocular surgery or ocular injury within 12 weeks of enrollment for this study.
* Anterior segment disease, infection, inflammation, or abnormality that contraindicates contact lens wear.
* History of herpetic keratitis.
* Slit-lamp findings at baseline as specified in the protocol.
* Any use of systemic or ocular medications for which contact lens wear could be contraindicated, including ocular medications that require instillation during contact lens wear.
* Clinically significant dry eye not responding to treatment.
* History of refractive surgery.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Nick, Dipl. Ing., Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 1 study center located in the US.
Pre-assignment Details: Of the 50 enrolled, 1 participant was exited as a screen failure prior to randomization and exposure to the study product. This reporting group includes all randomized participants (49).
Groups:
- Sequence 1: T1 and T2; T3 and T4; T5 and T6
- Sequence 2: T1 and T2; T5 and T6; T3 and T4
- Sequence 3: T3 and T4; T1 and T2; T5 and T6
- Sequence 4: T3 and T4; T5 and T6; T1 and T2
- Sequence 5: T5 and T6; T1 and T2; T3 and T4
- Sequence 6: T5 and T6; T3 and T4; T1 and T2
Period: Exposure Pair 1, 30 Minutes
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 8 | 8 | 8 | 8 | 8 | 9
Completed | 8 | 8 | 8 | 8 | 8 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Exposure Pair 2, 30 Minutes
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 8 | 8 | 8 | 8 | 8 | 9
Completed | 8 | 8 | 8 | 8 | 8 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Exposure Pair 3, 30 Minutes
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 8 | 8 | 8 | 8 | 8 | 9
Completed | 8 | 8 | 8 | 8 | 8 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects/eyes exposed to the investigational products (embossed or non-embossed lenses).
Groups:
- Overall: All treatment sequences
Arm/Group | Overall
Number analyzed (Participants) | 49
Age, Customized [Mean (Standard Deviation); unit: years]
  18 - 68 Years | 45.4 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Lenses With Axis Orientation ≤ 10 Degrees From Ideal Location After 3 Minutes of Wear
Description: Axis orientation (the rotational positioning of the lens on the eye) was indicated by an axis mark. The actual location of the axis mark was evaluated during slit lamp review and compared to the ideal location for the axis mark, with the difference measured in degrees (0 to +/- 180). The ideal location for the axis mark was iteration-specific (either 6 o'clock or 3 and 9 o'clock). This outcome measure was pre-specified for the embossed lenses only (TEST1, TEST3, and TEST5).
Time Frame: Day 1
Population: This analysis population includes all all randomized participants satisfying all of the inclusion/exclusion criteria.
Measure: Number; unit: percentage of lenses
Groups:
- TEST1: Iteration 2-87-1 with embossed mark
- TEST3: Iteration 2-87-2 with embossed mark
- TEST5: Iteration 2-87-3 with embossed mark
Arm/Group | TEST1 | TEST3 | TEST5
Number analyzed (Participants) | 49 | 49 | 49
percentage of lenses | 24.5 | 46.9 | 36.7

2. Secondary Outcome: Lens Awareness
Description: Lens awareness was assessed by the participant on a 5-point scale (0=none and 4=severe) within the first 5 minutes of wear for each eye separately.
Time Frame: Day 1
Population: This analysis population includes all all randomized participants satisfying all of the inclusion/exclusion criteria.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- TEST2: Iteration 2-87-1 without embossed mark
- TEST4: Iteration 2-87-2 without embossed mark
- TEST6: Iteration 2-87-3 without embossed mark
Arm/Group | TEST1 | TEST2 | TEST3 | TEST4 | TEST5 | TEST6
Number analyzed (Participants) | 49 | 49 | 49 | 49 | 49 | 49
units on a scale | 0.6 (0.8) | 0.2 (0.5) | 0.4 (0.7) | 0.2 (0.4) | 1.0 (1.1) | 0.6 (0.7)

3. Secondary Outcome: Handling on Removal
Description: Handling on removal (after 30 minutes of wear) was assessed by the participant on a scale from 1 to 10 (1=poor and 10=excellent). This outcome measure was pre-specified for the embossed lenses only (TEST1, TEST3, and TEST5).
Time Frame: Day 1
Population: This analysis population includes all all randomized participants satisfying all of the inclusion/exclusion criteria.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEST1 | TEST3 | TEST5
Number analyzed (Participants) | 49 | 49 | 49
units on a scale | 8.0 (2.4) | 7.8 (2.6) | 8.9 (1.8)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (18 days). This analysis group includes all participants/eyes exposed to the investigational products (embossed or non-embossed lenses).
Description: AEs were defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users, or other persons, whether or not related to the investigational medical device.
Groups:
- TEST (1,3,5): Delefilcon A toric contact lenses with embossed mark, 3 different iterations, crossover all on the same eye
- TEST (2,4,6): Delefilcon A toric contact lenses without embossed mark, 3 different iterations, crossover all on the same eye
Arm/Group | TEST (1,3,5) | TEST (2,4,6)
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 0/49 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No